CLINICAL TRIAL: NCT01499303
Title: Phase II Trial to Evaluate the Efficacy of Fostamatinib in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma(DLBCL)
Brief Title: Study to Learn if 200mg Test Drug (Fostamatinib) Helps People With Large B-Cell Lymphoma,a Type of Blood Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4302C00001
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: lymphoma; DLBCL; fostamatinib; Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — fostamatinib

ARMS (1):
- Fostamatinib 200 (Experimental): 200mg fostamatinib bid n=60
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Phase II Trial to evaluate the efficacy of 200mg fostamatinib

SUMMARY:
This study will evaluate the effectiveness of fostamatinib (200 mg twice a day) in patients with worsening or unmanageable lymphoma with a specific type of lymphoma called Diffuse Large B-Cell Lymphoma (abbreviated as DLBCL)

DETAILED DESCRIPTION:
Phase II Trial to Evaluate the Efficacy of Fostamatinib in Patients with Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years of age.
* Patients with relapsed or refractory diffuse large B-cell lymphoma who have previously received R-CHOP (or equivalent) chemo-immunotherapy and high dose chemotherapy with stem cell rescue, or who are ineligible for high dose therapy with stem cell rescue.
* Measurable disease as defined by Cheson et al 2007 criteria.
* One fresh pre-treatment excisional or core needle biopsy from suitable and accessible site.
* World Health Organization (WHO) performance status 0 to 1.

Exclusion Criteria:

* Treatment with nitrosurea, mitomycin C, investigational agents or study drugs w/in28 days of first dose of study treatment, any other chemotherapy, immunotherapy or anticancer agents w/in 3 weeks of first dose of study treatment, previous fostamatinib.
* With the exception of alopecia, any unresolved toxicities from prior therapy or surgery greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
* Uncontrolled hypertension (defined as >140mmHg systolic and/or > 90 mmHG diastolic at baseline with or without antihypertensive therapy.
* Evidence of tuberculosis (TB).
* Inadequate boen marrow reserve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Weidman, RN, MSN, PMP, Study Director — Sponsor GmbH
Locations (21):
- United States (19):
  - Research Site, Huntsville, Alabama
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Sarasota, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Iowa City, Iowa
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
- United Kingdom (2):
  - Research Site, London
  - Research Site, Southampton

REFERENCES:
- See also: D4302C00001_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1489&filename=D4302C00001_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the US and UK. Patient enrolment was completed on 14 June 2013. However three patients, considered by the Investigator to still be receiving clinical benefit, continue to receive fostamatinib. A total of 102 patients were enrolled and 68 received Fostamatinib doses of 100mg or 200mg and 38 Screen Failures.
Groups:
- 100mg BID: 100mg Fostmatinib BID
- 200mg BID: 200mg Fostmatinib BID
Period: Overall Study
Arm/Group | 100mg BID | 200mg BID
Started | 21 | 47
Completed | 18 | 40
Not Completed | 3 | 7
Not completed — Ongoing | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 4
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Most patients were male (69.1%). The mean age (± standard deviation) was 63.6 ± 12.6 years.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100mg BID | 200mg BID | Total
Number analyzed (Participants) | 21 | 47 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.38) | 63.9 (12.78) | 63.6 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 12 | 35 | 47

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Patients were assessed using the revised response criteria for malignant lymphoma (Cheson). Patients were assessed for response, with CT and FDG-PET scans at 8 weeks, then every 12 weeks until radiological progression by clinical CT. Complete response (CR) was defined as disappearance of all target and non-target lesions in the liver and spleen and all lymph node masses regressed to normal size. Partial response (PR) was defined as ≥50% reduction in sum of the product of the diameters (SPD) for measured lymph nodes, splenic and liver lesions separately compared to baseline SPD. Objective response rate (CR + PR) analysis, exact binomial test, primary analysis.
Time Frame: Week 8
Population: Full analysis set - all randomised patients
Measure: Number (95% Confidence Interval); unit: Patients
Arm/Group | 100mg BID | 200mg BID
Number analyzed (Participants) | 21 | 47
Patients | 2 [1.17 to 30.38] | 0 [0.00 to 7.55]

ADVERSE EVENTS:
Arm/Group | 100mg BID | 200mg BID
Serious Adverse Events (participants affected / at risk) | 3/21 | 12/47
Other Adverse Events (participants affected / at risk) | 21/21 | 44/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100mg BID (N=21) | 200mg BID (N=47)
PNEUMONIA (Infections and infestations) | 0 | 2
CELLULITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 1
FATIGUE (General disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100mg BID (N=21) | 200mg BID (N=47)
DIARRHOEA (Gastrointestinal disorders) | 3 | 16
CONSTIPATION (Gastrointestinal disorders) | 4 | 12
NAUSEA (Gastrointestinal disorders) | 4 | 12
VOMITING (Gastrointestinal disorders) | 0 | 9
FATIGUE (General disorders) | 4 | 13
PYREXIA (General disorders) | 4 | 10
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 8
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 | 5
BLOOD CREATININE INCREASED (Investigations) | 3 | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 3 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 12
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
HYPERTENSION (Vascular disorders) | 1 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 5
HEADACHE (Nervous system disorders) | 2 | 5
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 4
OEDEMA PERIPHERAL (General disorders) | 2 | 3
ASTHENIA (General disorders) | 0 | 3
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 3
BLOOD UREA INCREASED (Investigations) | 2 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0
HYPOTENSION (Vascular disorders) | 2 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3
SYNCOPE (Nervous system disorders) | 0 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 4
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 4
PNEUMONIA (Infections and infestations) | 0 | 3
ANXIETY (Psychiatric disorders) | 2 | 4
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No